CLINICAL TRIAL: NCT04384458
Title: Comparative Study of Hydroxychloroquine and Ivermectin in COVID-19 Prophylaxis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara (Other)
Responsible Party: Principal Investigator, betemora, MD, PhD, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCQ+IVM
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Coronavirus Infections
Keywords: Coronavirus Infections; Health Personnel; Hydroxychloroquine; Pre-Exposure Prophylaxis; Antimalarials; Antirheumatic Agents; Ivermectin
MeSH Terms: conditions — Coronavirus Infections | interventions — Hydroxychloroquine; Ivermectin

STUDY DESIGN:
Intervention Model Description: The study is a open-blind, randomised trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Active Comparator): Oral hydroxychloroquine 400 mg twice a day on day 1, one 400 mg tablet on day 2, 3, 4, and 5, followed by one 400 mg tablets every 05 days until day 50th associated with with 20 milligrams twice on day of active zinc for 45 consecutive days
  Interventions: Drug: Hydroxychloroquine
- Ivermectin (Active Comparator): Oral ivermectin dosage guidelines based on participant body weight, once on day for 2 consecutive days. This dose schedule should be repeated every 14 days for 45 days associated with 20 milligrams twice on day of active zinc.
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Hydroxychloroquine — Oral hydroxychloroquine 400 mg twice a day on day 1, one 400 mg tablet on day 2, 3, 4, and 5, followed by one 400 mg tablets every 05 days until day 50th associated with 66 mg of zinc sulfate.
  Arms: Hydroxychloroquine
Drug: Ivermectin — Oral ivermectin dosage guidelines based on participant body weight, once on day for 2 consecutive days. This dose schedule should be repeated every 14 days for 45 days associated with 20 milligrams twice on day of active zinc.
  Arms: Ivermectin

SUMMARY:
We have to be aware of the challenge and concerns brought by 2019-nCoV to our healthcare workers. Front-line healthcare workers can become infected in the management of patients with COVID-19; the high viral load in the atmosphere, and infected medical equipment are sources for the spread of SARS-CoV-2. If prevention and control measures are not in place, these healthcare workers are at great risk of infection and become the inadvertent carriers to patients who are in hospital for other diseases. Nowadays a question that has not yet been clarified by science has been arises: is hydroxychloroquine associated with zinc compared to ivermectin associated with zinc effective as a prophylaxis for asymptomatic professionals involved in the treatment of suspected or confirmed case of COVID-19?

DETAILED DESCRIPTION:
The study is a open-blind, randomised trial that will be conducted in asymptomatic professionals working in areas of high exposure and high risk of transmission of SARS-COV-2.

After obtaining fully informed consent, the investigator will recruit workers in areas of high exposure and high risk of transmission of SARS-COV-2.

Participants will be divided into 2 groups:

* Hydroxychloroquine (HCQ) = 400mg twice on day 1, 400mg/day on day 2, 3, 4, and 5 followed by 400mg once every 05 days, for the next 7 weeks associated with 20 milligrams twice on day of active zinc for 45 consecutive days;
* Ivermectin (IVM) = Dosage guidelines based on participant body weight, once on day for 2 consecutive days, This dose schedule should be repeated every 14 days for 45 days associated with 20 milligrams twice on day of active zinc.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 70 years;
* Professionals working in areas of high exposure and high risk of transmission of SARS-COV-2;
* Understands and agrees to comply with planned study procedures;
* Signed informed consent for participation in the study.

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Major allergy to Hidroxychloroquine, chloroquine or 4-aminoquinolines;
* Serum potassium lower than 3.4 mEq/l;
* Serum magnesium lower than 1.7 mg/dL;
* QTc interval > 470 ms for man and > 480 ms for woman;
* Weight < 40 kg;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants in whom there was a positivity for SARS-CoV-2. | Post-intervention at day 52
  Proportion of participants in whom there was a a positivity for SARS-CoV-2 through specific examination (RT-PCR) or by serology for antibodies specific (IgM and IgG), corroborated or not with clinical finding of COVID-19, defined as the occurrence of signs and symptoms suggestive of this disease.

SECONDARY OUTCOMES:
Participants who developed mild, moderate, or severe forms of COVID-19. | Post-intervention at day 52.
  Proportion of participants who developed mild, moderate, or severe forms of COVID-19.
Measurement of the QT interval. | Baseline, 3, 15 and 45 days post-intervention.
  Measurement of the QT interval through electrocardiogram evaluation.
Widening of the corrected QT interval or with changes in heart rate on the ECG. | Day 52.
  Proportion of participants who evolved with widening of the corrected QT interval or with changes in heart rate on the ECG.
Comparison of hematological and biochemical parameters. | Day 52.
  Comparison of baseline (visit 0) and final (visit 5) values of hematological and biochemical parameters.
Occurrence of adverse events. | Post-intervention at day 52.
  Proportion of occurrence of adverse events reported by participants or verified by the attending physician, or even observed in laboratory tests.
Assessment of COVID-19 symptom severity. | Post-intervention at day 52.
  Severity of symptoms of COVID-19 measured by a visual analog scale (VAS), with scores ranging from zero to 10, where zero represents the absence of the symptom and 10 corresponds to the most intense manifestation of symptoms (severe dyspnoea).
Proportion of participants who discontinue study intervention. | Post-intervention at day 52.
  Proportion of participants who discontinue study intervention,
Proportion of participants who required hospital care. | Post-intervention at day 52.
  Proportion of participants who required hospital care.
Proportion of participants who required mechanical ventilation. | Post-intervention at day 52.
  Proportion of participants who required mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Drug Research and Development Center (NPDM), Federal University of Ceará (UFC), Fortaleza, Ceará, Brazil